CLINICAL TRIAL: NCT06140160
Title: Anterior Thoracic Perforating Artery (PATA); Systematization and Applications in Reconstructive Surgery of the Head and Neck
Acronym: PATA-Fix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: mermoz hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-A00784-41
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Upper Aero-intestinal Tract Cancer; Supraclavicular Flap; Anterior Thoracic Perforator Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with an indication for Doppler ultrasound of the supra-aortic trunks (Experimental)
  Interventions: Procedure: Doppler ultrasound

INTERVENTIONS:
Procedure: Doppler ultrasound — To carry out an additional measurement using Doppler ultrasound (non-invasive examination). Doppler ultrasound measurements of the diameter and length of the perforating artery using a high-frequency Doppler ultrasound probe following a Doppler ultrasound of the supra-aortic trunks.

SUMMARY:
The use of cutaneous or fasciocutaneous flaps is daily in reconstructive surgery ENT in patients with cancers of the upper aero-digestive tract (AVDS). Cancers of the oral cavity require reconstructions with thin flaps in order to best preserve the functions of swallowing and phonation via patients' joints. Indeed, the flaps are inert tissues, which can only be mobilized by the residual muscles of the patients' tongue: their lightness and finesse facilitates this mobilization. The use of free flaps is regular but requires micro-surgical skill of the operator as well as a preserved general condition of the patients and appropriate post-operative care. Alternatively, there are some pedicled flaps with the appropriate thickness to reconstruct extensive loss of substances from the oral cavity in a suitable manner: the supraclavicular flap, the suprahyoid flap, the submental flap and the myo-mucosal flap pedicled on the facial artery being more limited in size. The creation of an anterior thoracic fasciocutaneous flap, pedicled on the anterior thoracic perforating artery (PATA) seems to be another suitable therapeutic option. Only one preliminary Chinese study describes it, on only eleven patients. According to the authors, it would offer a wide skin palette (up to 15x10cm). Its long pedicle (on average 9.2cm) would allow a significant axis of rotation so that the flap easily reaches the oral cavity. The authors underline the variability of the origin of this perforator, arising depending on the case from the transverse cervical trunk (9 cases) or from the supraclavicular artery (2 cases), branches of division of the thyro-cervical trunk.

However, when the PATA arises from the supraclavicular artery, its interest could be limited because the creation of a PATA perforator flap could compromise the creation of a secondary supraclavicular flap.

Thus, this study aims to clarify the feasibility of harvesting the PATA flap in the greatest number of patients. The objective is to study the variations of the anterior thoracic perforating artery necessary for the creation of this flap, by specifying its vascularization territory and its characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patient, man or woman over 18 years old,
* Patient admitted for an indication for Doppler ultrasound of the supra-aortic trunks (previously prescribed for any medical reason),
* Patient having received written information and collection of the non-opposition of the patient to participate in the study,
* Patient affiliated or beneficiary of a security regime social.

Exclusion Criteria:

* Minor patient,
* History of cervical surgery,
* Patients who have an inaccessible morphology to an exploration of the lower lateral cervical region, high, below and above the right and left clavicle such as the small necks, and/or with dermato-sclerosis,
* Patients who do not have the intellectual or physical allowing them to give their consent,
* Patient in period of exclusion due to another research still in progress at the time of inclusion,
* Refusal to participate in the patient's study,
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial decision or administrative,
* Pregnant, breastfeeding or parturient woman,
* Patient hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-03-19 (Estimated); Study Completion 2024-09-19 (Estimated)

PRIMARY OUTCOMES:
Existence of the anterior thoracic perforating artery | 1 hour
  existence of the anterior thoracic perforating artery (PATA) : yes/no
Presence of the anterior thoracic perforating artery | 1 hour
  the presence of the anterior thoracic perforating artery on the left and right,
Origin of anterior thoracic perforating artery | 1 hour
  Origin of anterior thoracic perforating artery : transverse cervical trunk/ supraclavicular artery

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France